CLINICAL TRIAL: NCT04572165
Title: Epidemiological Assessment of the Risk for Pancreatic Cancer Associated With the Use of Semaglutide in Patients With Type 2 Diabetes - A Cohort Study Based on Nordic Registry Data
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Novo Nordisk A/S (Industry)
Collaborators: Department of Public Health, University of Southern Denmark (Unknown)
Responsible Party: Sponsor
Other Study IDs: NN9535-4447; U1111-1214-6228 (Other: World Health Organization (WHO)); EUPAS37258 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2020-09-30; First posted 2020-10-01 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- semaglutide: New users of Ozempic® or Rybelsus®
  Interventions: Drug: Ozempic®; Drug: Rybelsus®
- Active comparator: First-time ever users of an active comparator drug
  Interventions: Drug: Active Comparator

INTERVENTIONS:
Drug: Ozempic® — Patients have been treated with commercially available Ozempic® according to local label and to routine clinical practice at the discretion of the treating physician. The decision to initiate treatment with commercially available Ozempic® had been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before and independently from the decision to include the patient in this study.
  Groups: semaglutide
Drug: Active Comparator — Patients have been treated with commercially available active comparators according to local label and to routine clinical practice at the discretion of the treating physician. Active comparators will include the following antidiabetic agents: sulphonylureas, sodium-glucose co-transporter 2 inhibitors, and insulin. The decision to initiate treatment with commercially available active comparators had been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before and independently from the decision to include the patient in this study.
  Groups: Active comparator
Drug: Rybelsus® — Patients have been treated with commercially available Rybelsus® according to local label and to routine clinical practice at the discretion of the treating physician. The decision to initiate treatment with commercially available Rybelsus® had been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before and independently from the decision to include the patient in this study.
  Groups: semaglutide

SUMMARY:
The aim of this study is to evaluate whether exposure to semaglutide influences the risk of pancreatic cancer in patients with type 2 diabetes. This is achieved by estimating the risk of pancreatic cancer associated with semaglutide use as compared to use of other non-incretin antidiabetic drugs used at a similar stage as Ozempic® or Rybelsus® in the treatment of type 2 diabetes. A multi-national, non-interventional study based on health care data from Denmark, Sweden, and Norway is conducted covering the period 2018-2023. A cohort study design is used comparing new users of semaglutide with new users of other antidiabetic drugs used at a similar stage as Ozempic® or Rybelsus® in the treatment of type 2 diabetes (active comparators). Active comparators will include the following non-incretin antidiabetic agents: sulphonylureas, sodium-glucose co-transporter 2 inhibitors, and insulin subdivided into i) basal insulin only and ii) basal + bolus insulin or premix insulin. Propensity scores are used to match new users of semaglutide with new users of active comparators. National prescription-, cancer- and patient registries are used to identify exposure to antidiabetic agents, pancreatic cancer cases, and covariates to be used in propensity score matching. This study is a post-authorisation safety study (PASS).

ELIGIBILITY:
Inclusion Criteria:

* Use of semaglutide or initiation of active comparators from when the first subject is dispensed semaglutide in the respective country (2018) until December 31, 2022. Initiation is defined as no previous prescription of a drug with the same active ingredient in the past 10 years as recorded in the national prescription registries. Previous use of the same class of drug is however accepted. Further, a patient who shift from Ozempic® to Rybelsus® or vice versa will be considered a continued user in the semaglutide group.
* At least two prescriptions of either semaglutide or active comparators (at the level of the active ingredient) with the second prescription filled less than one year after the initial prescription. Two prescriptions filled at first day of treatment will, however, only be counted as one prescription.
* 18 years or older at the cohort entry date. The cohort entry date is defined as the dispensing date of the initial prescription (i.e. treatment initiation).
* Ten years or more of continuous residency in the country of residence before initiation of semaglutide or active comparators.

Exclusion Criteria:

Patients with rare but strong risk factors for developing pancreatic cancer are excluded. Therefore, patients with any history of the following conditions (identified according to 10th version of International Classification of Diseases [ICD-10]) before cohort entry date (based on the last 10 years of data or more) are excluded:

* A history of any cancer except non-melanoma skin cancer
* Acute pancreatitis
* Alcohol-induced chronic pancreatitis
* Other chronic pancreatitis
* Cystic fibrosis
* Other phacomatoses, not elsewhere classified (including Peutz-Jeghers syndrome and Von Hippel-Lindau syndrome)
* Neurofibromatosis (non-malignant, Von Recklinghausen disease)

In addition, the following patients are excluded:

* Patients with a history of pancreatic cancer as these patients are no longer at risk for an incident pancreatic cancer
* Patients who initially started insulin as first-line antidiabetic treatment and who did not add on or switch to non-insulin treatment within 3 months. Those initiating insulin as first-line treatment during the study period is disregarded in terms of study inclusion, although they may be included upon initiating additional therapy, provided it is started within three months.
* Patients with polycystic ovary syndrome (PCOS)
* Patients with gestational diabetes
* Patients who meet one of the conditions used as exclusion criteria listed above (except acute and chronic pancreatitis) after cohort entry date but before start of follow-up (i.e. during the first year after treatment initiation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The risk of pancreatic cancer is compared in a cohort of first-time ever users of semaglutide relative to a cohort of first-time ever users of the other antidiabetic drugs used at a similar stage as Ozempic® or Rybelsus® in the treatment of type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 600000 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of first time malignant neoplasm of pancreas | From when semaglutide entered the market in Denmark, Sweden, and Norway (Q3/Q4 2018) until December 31, 2023
  Incidence

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com